CLINICAL TRIAL: NCT05853159
Title: Clinical and Radiological Prognostic Factors of Acute Necrotizing Encephalopathy in Sohag University Hospital
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Marwa Mahmoud Fathy, Pediatric and Neonatology Resident at Sohag University Hospital, Sohag University
Other Study IDs: Soh-med-23-04-07-MS
Record Dates: First submitted 2023-04-19; First posted 2023-05-10 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Acute Necrotizing Encephalopathy
MeSH Terms: conditions — Leukoencephalitis, Acute Hemorrhagic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Basic Laboratory investigations , Cerebrospinal fluid analysis — to detect severity and prognostic factors of Acute Necrotizing Encephalopathy
  Other Names: MRI brain

SUMMARY:
Acute necrotizing encephalopathy of childhood (ANEC) is a fulminant type of encephalopathy. Most reported cases occur in Asian children with the highest prevalence among patients between the age of 6 and 18 months. The most common clinical presentations are fever, rapid alteration in the level of consciousness, and seizures, in addition to characteristic findings in brain imaging that include, but are not limited to, bilateral thalamic lesions with supra and infra-tentorial lesions of variable dimensions.

The diagnosis of ANEC was determined by specific diagnostic criteria as described by Mizuguchi [1] which consist of

1. Encephalopathy preceded by viral febrile illness with rapid deterioration in the level of consciousness and convulsions.
2. Absent cerebrospinal fluid (CSF) pleocytosis.
3. Symmetric multifocal brain lesions.
4. Elevation in serum aminotransferase levels.
5. Exclusion of similar diseases. The ANE severity score was used to assess the severity of illness after admission for shock (3 points), brainstem lesions (2 points), age >4 years (2 points), platelet (PLT) count < 100,000 (1 point), and elevated CSF protein (1 point) was observed. [3] A total score of 9

ELIGIBILITY:
Inclusion Criteria:

- Children aged from 2months up to 12 years admitted to the pediatric emergency department or pediatric ICU presented with Acute encephalopathy & meet diagnostic criteria of acute necrotizing encephalopathy or come for follow up in our outpatient clinic.

Exclusion Criteria:

* Children known to have metabolic disease. Children who have picture of CNS infection & confirmed by CSF analysis.

Ages: 2 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged from 2months up to 12 years admitted to the pediatric emergency department or pediatric ICU presented with Acute encephalopathy & meet diagnostic criteria of acute necrotizing encephalopathy or come for follow up in our outpatient clinic.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Acute necrotizing encephalitis severity score | one year
  Clinical and Radiological Prognostic Factors of Acute Necrotizing Encephalopathy in Sohag University Hospital

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bashiri FA, Al Johani S, Hamad MH, Kentab AY, Alwadei AH, Hundallah K, Hasan HH, Alshuaibi W, Jad L, Alrifai MT, Hudairi A, Al Sheikh R, Alenizi A, Alharthi NA, Abdelmagid TA, Ba-Armah D, Salih MA, Tabarki B. Acute Necrotizing Encephalopathy of Childhood: A Multicenter Experience in Saudi Arabia. Front Pediatr. 2020 Oct 9;8:526. doi: 10.3389/fped.2020.00526. eCollection 2020. PMID 33163461
- [Background] Levine JM, Ahsan N, Ho E, Santoro JD. Genetic Acute Necrotizing Encephalopathy Associated with RANBP2: Clinical and Therapeutic Implications in Pediatrics. Mult Scler Relat Disord. 2020 Aug;43:102194. doi: 10.1016/j.msard.2020.102194. Epub 2020 May 15. PMID 32426208
- [Background] Wu L, Peng H, Jiang Y, He L, Jiang L, Hu Y. Clinical features and imaging manifestations of acute necrotizing encephalopathy in children. Int J Dev Neurosci. 2022 Aug;82(5):447-457. doi: 10.1002/jdn.10201. Epub 2022 Jun 22. PMID 35688614
- [Background] Song Y, Li S, Xiao W, Shen J, Ma W, Wang Q, Yang H, Liu G, Hong Y, Li P, Yang S. Influenza-Associated Encephalopathy and Acute Necrotizing Encephalopathy in Children: A Retrospective Single-Center Study. Med Sci Monit. 2021 Jan 3;27:e928374. doi: 10.12659/MSM.928374. PMID 33388740